CLINICAL TRIAL: NCT00557024
Title: Radiotherapy as an Adjuvant Therapy After Radiofrequency Ablation for Hepatocellular Carcinoma
Acronym: RT-RFA
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: cancer canter, Sun Yat-sen University, cancer canter, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: rfa-004
Record Dates: First submitted 2007-11-09; First posted 2007-11-12 (Estimated); Last update posted 2008-11-18 (Estimated); Status verified 2008-11

CONDITIONS: Hepatocellular Carcinoma; Liver Cancer
Keywords: hepatocellular carcinoma; liver cancer; radiofrequency ablation; radiotherapy; adjuvant therapy
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): radiotherapy after RFA
  Interventions: Procedure: radiotherapy after RFA
- 2 (Active Comparator): RFA alone
  Interventions: Procedure: RFA

INTERVENTIONS:
Procedure: RFA — radiofrequency ablation
  Arms: 2
Procedure: radiotherapy after RFA — radiotherapy after RFA
  Other Names: RT-RFA
  Arms: 1

SUMMARY:
The purpose of the investigators study is to prospectively evaluate whether radiotherapy as an adjuvant therapy after RFA will improve the outcome of radiofrequency ablation for hepatocellular carcinoma (HCC) or not.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 - 75 years, who refused surgery
* A solitary HCC ≤ 7.0cm in diameter, or multiple HCC ≤ 3 lesions, each ≤ 3.0cm in diameter
* Lesions being visible on ultrasound (US) and with an acceptable/safe path between the lesion and the skin as shown on US,
* No extrahepatic metastasis
* No imaging evidence of invasion into the major portal/hepatic vein branches
* No history of encephalopathy, ascites refractory to diuretics or variceal bleeding
* A platelet count of > 40,000/mm3
* No previous treatment of HCC except liver resection.

Exclusion Criteria:

* Patient compliance is poor
* The blood supply of tumor lesions is absolutely poor or arterial-venous shunt that TACE can not be performed
* Previous or concurrent cancer that is distinct in primary site or histology from HCC, EXCEPT cervical carcinoma in situ, treated basal cell carcinoma, superficial bladder tumors (Ta, Tis & T1). Any cancer curatively treated > 3 years prior to entry is permitted.
* History of cardiac disease:

  * congestive heart failure > New York Heart Association (NYHA) class 2;
  * active coronary artery disease (myocardial infarction more than 6 months prior to study entry is permitted);
  * cardiac arrhythmias requiring anti-arrhythmic therapy other than beta blockers, calcium channel blocker or digoxin; or
  * uncontrolled hypertension (failure of diastolic blood pressure to fall below 90 mmHg, despite the use of 3 antihypertensive drugs).
* Active clinically serious infections ( > grade 2 National Cancer Institute [NCI]-Common Terminology Criteria for Adverse Events [CTCAE] version 3.0)
* Known history of human immunodeficiency virus (HIV) infection
* Known Central Nervous System tumors including metastatic brain disease
* Patients with clinically significant gastrointestinal bleeding within 30 days prior to study entry
* Distantly extrahepatic metastasis
* History of organ allograft
* Substance abuse, medical, psychological or social conditions that may interfere with the patient's participation in the study or evaluation of the study results
* Known or suspected allergy to the investigational agent or any agent given in association with this trial
* Any condition that is unstable or which could jeopardize the safety of the patient and his/her compliance in the study
* Pregnant or breast-feeding patients. Women of childbearing potential must have a negative pregnancy test performed within seven days prior to the start of study drug. Both men and women enrolled in this trial must use adequate barrier birth control measures during the course of the trial.
* Excluded therapies and medications, previous and concomitant:

  * Prior use of any systemic anti-cancer treatment for HCC, eg. chemotherapy, immunotherapy or hormonal therapy (except that hormonal therapy for supportive care is permitted). Antiviral treatment is allowed, however interferon therapy must be stopped at least 4 weeks prior randomization.
  * Prior use of systemic investigational agents for HCC
  * Autologous bone marrow transplant or stem cell rescue within four months of start of study drug

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2007-11; Primary Completion 2009-11 (Estimated); Study Completion 2010-07 (Estimated)

PRIMARY OUTCOMES:
Overall survivals | 3, abd 5-years

SECONDARY OUTCOMES:
Recurrence rates | 3-, and 5-years

CONTACTS AND LOCATIONS:
Overall Officials: min-shan chen, doctor, Principal Investigator — Department of Hepatobilliary Surgery, Cancer Center, Sun Yat-sen University
Locations (1):
- Department of Hepatobilliary Surgery, Cancer Center, Sun Yat-sen University, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Poon RT, Fan ST, Tsang FH, Wong J. Locoregional therapies for hepatocellular carcinoma: a critical review from the surgeon's perspective. Ann Surg. 2002 Apr;235(4):466-86. doi: 10.1097/00000658-200204000-00004. PMID 11923602
- [Background] Chen MS, Li JQ, Zheng Y, Guo RP, Liang HH, Zhang YQ, Lin XJ, Lau WY. A prospective randomized trial comparing percutaneous local ablative therapy and partial hepatectomy for small hepatocellular carcinoma. Ann Surg. 2006 Mar;243(3):321-8. doi: 10.1097/01.sla.0000201480.65519.b8. PMID 16495695
- [Background] Buscarini L, Buscarini E, Di Stasi M, Vallisa D, Quaretti P, Rocca A. Percutaneous radiofrequency ablation of small hepatocellular carcinoma: long-term results. Eur Radiol. 2001;11(6):914-21. doi: 10.1007/s003300000659. PMID 11419162